CLINICAL TRIAL: NCT00572429
Title: Effects of Mixed Exercise Regime and L-Carnitine Supplementation on Kinetics of Triglyceride-rich Lipoproteins in HIV Patients on HAART
Brief Title: Effects of Mixed Exercise Regime and L-Carnitine Supplementation in HIV Patients on HAART
Acronym: HIV
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subjects enrolled,study never started
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 200715081
Record Dates: First submitted 2007-12-11; First posted 2007-12-13 (Estimated); Last update posted 2012-12-19 (Estimated); Status verified 2012-12

CONDITIONS: HIV Infections; Hyperlipidemia; Exercise
Keywords: HIV/AIDS; HAART; high cholesterol; exercise; L-carnitine; Complimentary therapies
MeSH Terms: conditions — HIV Infections; Hyperlipidemias; Motor Activity; Acquired Immunodeficiency Syndrome; Hypercholesterolemia | interventions — Carnitine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Placebo Comparator)
  Interventions: Dietary Supplement: l-carnitine

INTERVENTIONS:
Dietary Supplement: l-carnitine — 3 gram daily dose

SUMMARY:
HIV patients treated with Highly Active AntiRetroviral Therapy (HAART) show significant metabolic symptoms, such as lipodystrophy, dyslipidemia, and insulin resistance. A possible contribution to these symptoms in HIV/HAART is a decrease in mitochondrial function, resulting in a decreased fatty acid oxidation. A combined regime of aerobic and resistance training has been demonstrated to increase lean body mass and reduce overall fat and truncal fat and the levels of triglyceride and LDL cholesterol.

DETAILED DESCRIPTION:
The introduction of Highly Active AntiRetroviral Therapy (HAART) for AIDS and HIV has improved survival considerably. However, HIV patients treated with HAART show significant metabolic symptoms, such as lipodystrophy, dyslipidemia, and insulin resistance. A possible contribution to these dysmetabolic symptoms in HIV/HAART is a decrease in mitochondrial function, resulting in a decreased fatty acid oxidation. Life style modulation such as aerobic exercise and L-carnitine supplementation may be beneficial to mitochondrial function. Aerobic exercise improves the biogenesis and function of mitochondria. A combined regime of aerobic and resistance training has been demonstrated to increase lean body mass and reduce overall fat and truncal fat and the levels of triglyceride and LDL cholesterol. L-Carnitine plays an important role in the transfer of long-chain acyl groups into the mitochondrial matrix and potentially improves energy metabolism. Further, L-carnitine supplementation decreases serum triglyceride levels in HIV/HAART patients with hypertriglyceridemia. However, little is known whether these life style modulations act synergistically in HIV/HAART patients.

We hypothesize that a mixed regimen of exercise (including both resistance and aerobic exercise) and L-carnitine supplementation will improve mitochondrial dysfunction in HIV/HAART patients, and therefore, alleviate dysmetabolic symptoms such as dyslipidemia and insulin resistance. In this randomized, placebo-controlled study, we will explore whether a mixed regimen of exercise, including both resistance and aerobic exercise, and L-carnitine supplementation affect lipids and remnant lipoproteins, adipokines, insulin resistance; blood lactate levels and VO2max; and kinetics of leucine and triglyceride-rich lipoproteins among African-American and Hispanic HIV-positive subjects undergoing HAART. Effects on muscle mitochondrial function will be assessed using exercise tests and body composition assessment (DEXA and Bioimpedance), while effects on hepatic mitochondrial function will be assessed measuring the relation between leucine and VLDL-apoB metabolism. We believe that the proposed study will help to elucidate underlying mechanisms for metabolic complications and will offer new possibilities for intervention to reduce negative metabolic effects in HIV/HAART patients.

ELIGIBILITY:
Inclusion Criteria:

* African American, Hispanic and Caucasian adults with HIV on a stable HAART regimen (either PI or NNRTI based) for at least the past 6 months between 18 to 70 years of age.
* Patients taking SSRI's (Selective Serotonin Reuptake Inhibitors), SNRI's (Serotonin/Norepinephrine Reuptake inhibitors) and Tetracyclic antidepressants will be included as the risk of seizure in these patients in combination with the L-Carnitine supplement would be rare. Patients on these medications should be on a stable dose for at least 4-6 months prior to enrollment in the study.

Exclusion Criteria:

* Diabetes Mellitus
* Cushing's syndrome
* Renal disease (i.e. CKD Stages 3-5)
* Unstable liver disease
* Untreated thyroid dysfunction
* Seizure disorder
* Patients with conditions that can lower seizure threshold (i.e. brain tumors) or are taking medication(s) known to lower seizure threshold
* Pregnant or nursing mothers
* BMI > 35
* Ongoing hormone replacement therapy
* Hemoglobin levels less than 11 g/dl, and fasting triglyceride levels > 500 mg/dl.
* Subjects with ongoing hypolipidemic and warfarin therapy will be excluded. Additionally, patients taking Valproic Acid and / or Zidovudine will be excluded as these have been shown to deplete carnitine.
* Patients taking Venlafaxine and Bupropion will be excluded as these medications have a small risk (0.26% and 0.1-0.4% risk, respectively) of causing seizure in patients without a previous risk of seizure.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Exercise and L-carnitine supplementation will reduce blood lactate levels, increase the VO2sub-max and the VLDL to leucine enrichment ratio in HIV/HAART patients, suggesting an overall improvement of muscle and hepatic mitochondrial function. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lars Berglund, MD, PhD, Principal Investigator — UC Davis Health System
Locations (1):
- CARES, Sacramento, California, United States